CLINICAL TRIAL: NCT06917781
Title: Prostate Cancer Burden and Heterogeneity Evaluation Towards Liquid Biopsy: a Correlation Study to 18FDCFPyL PET and Patients Outcome
Acronym: TAYLOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25GENH01
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; 18F-PET-PSMA; Circulating Tumor Cells; Liquid biopsy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with prostate cancer (Other)
  Interventions: Other: Patients with 18F-PET-PSMA indication

INTERVENTIONS:
Other: Patients with 18F-PET-PSMA indication — Blood samples taken on several occasions:
  * before the 18F-PSMA PET scan for extension assessment, for all patients.
  * at 2nd and 4th treatment cycles (prior to treatment administration), only for patients receiving PLUVICTO® therapy.
  During the 1st treatment cycle, samples (optional for the patient) may also be taken at 5 different post-perfusion times.
  In addition, all imaging examinations performed during the study (standard 18F-PSMA PET scans) will be collected and centralized by the Sponsor for analysis.

SUMMARY:
This is a prospective, monocentric, proof of concept study aims to identify in prostate cancer patients, a potential relationship between CTC-PSMA positivity and 18F-PET-PSMA results as well as patient outcome.

Patients with 18F-PET-PSMA indication will perform imaging extension work-up as part of current practice. If they agree to participate in the study, a blood sample will be performed prior to the 18F-PET-PSMA standard imaging (T1).

In order to evaluate the potential relationship between CTC-PSMA and 18F-PET-PSMA imaging, the study will be presented to all patients seen in consultation for an extension workup for prostate cancer. This will allow to analyze the results in patients with different level of tumor burden afterward to define the following three groups based on imaging results:

Group 1 : no tumor volume Negative 18F-PET-PSMA (patients without uptake lesion)

Group 2 : low or medium tumor volume Positive 18F-PET-PSMA (patients with an uptake in prostate bed or with an oligo-metastatic extension (number of lesions < 6))

Group 3 : high tumor volume Positive 18F-PET-PSMA (patients with a polymetastastatic extension (number of lesions ≥ 6)).

In each of these groups, the rate of patients with positive PSMA CTC will be analyzed (i.e. patient having at least one CTC-PSMA positive).

For patients with an indication of treatment by 177LuPSMA-617 (PLUVICTO®) according to standard practices, additional blood samples will also be collected at the following time points: 2nd cycle (T2) and 4th cycle of treatment (T3), just before injection. For these patients, data will be collected up to 6 months after the last treatment injection (clinical and biological data; results of tumor assessments based on 18F-PET-PSMA imaging).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically confirmed adenocarcinoma of the prostate
3. Indication for 18F-PET-PSMA imaging
4. Signed written informed consent
5. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol
6. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Patients with a contraindication to 18F-PET-PSMA
2. Patient with an established neuro endocrine prostate cancer
3. Concurrent malignancy known to express a significant amount of PSMA (renal cancer, salivary gland tumors)
4. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
5. Patient who has forfeited his freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
The rate of patients presenting at least one (i.e >0) CTC-PSMA positive. | 1 day for each patient
  The rate of patients presenting at least one CTC-PSMA positive is defined as the ratio of the number of patients having at least one CTC-PSMA positive divided by the total number of patients evaluable in each group (G1, G2, G3).

SECONDARY OUTCOMES:
The number of CTC-PSMA positive will be evaluated at inclusion for each group and just before the 2nd and 4th course of 177LuPSMA (C2/C4). | 18 weeks for each patient
CTC-PSMA change will be defined as the number of CTC-PSMA positive at C2/C4 minus the number of CTC-PSMA positive at inclusion, if feasible. | 18 weeks for each patient
The total number of CTC will be evaluated. | 18 weeks for each patient
The response to 177LuPSMA | 15 months
  It will be evaluated according to investigator judgement and PSMA uptake alteration on PET as proposed in PROMISE V2.

CONTACTS AND LOCATIONS:
Locations (1):
- IUCT-O, Toulouse, France